CLINICAL TRIAL: NCT03100695
Title: A Prospective, Randomised, Single-centre Feasibility Study of Combined Autologous Platelet-rich Plasma and Concentrated Autologous Bone Marrow in Adult Patients With a Fresh Unilateral Tibial Diaphyseal Fracture Treated With Either Fine Wire Ring Fixator Device (Ilizarov) or Reamed Intramedullary Nailing
Brief Title: Tibial Fracture - Platelet-rich Plasma and Bone Marrow Concentrate
Acronym: T-PAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, PeterGiannoudis, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 226136
Record Dates: First submitted 2017-03-20; First posted 2017-04-04 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Unilateral Tibial Diaphyseal Fracture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients will undergo operative procedure with no additional intervention.
- Study (Experimental): Patients will undergo usual operative procedure with the addition of an injection of autologous, concentrated PRP-BMA at the site of fixation.
  Interventions: Other: Concentrated autologous PRP-BMA

INTERVENTIONS:
Other: Concentrated autologous PRP-BMA — Injection of autologous, concentrated platelet-rich plasma and bone marrow aspirate at the site of fixation.
  Arms: Study

SUMMARY:
A prospective, randomised study is to investigate the feasibility of conducting a superiority randomised controlled trial comparing the application of combined autologous PRP and concentrated autologous bone marrow (PRP-BMA) in addition to standard of care (either reamed intramedullary nailing or fine wire ring external fixator) for patients presenting with fresh tibial diaphyseal fractures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65, skeletally mature adults.
* Acute unilateral closed tibia diaphyseal fractures as the primary injury.
* Definitive fracture fixation with reamed intramedullary nailing (statically locked) or fine wire ring external fixator to be performed within 14 days from the date of injury.
* Willing and able (in the opinion of the study team) to provide informed consent and participate in all study activities.

Exclusion Criteria:

* Open/compound tibial fracture.
* Fracture Type 42-C2 according to Muller AO classification.
* Multi-segmental nature of this fracture (more than one fracture site within tibia for intervention.)
* Polytrauma (defined as injury severity score of 17 or more.)
* Prior or concomitant illnesses that may affect healing.
* Exposure to drugs that can affect the bone metabolic state within the past three months.
* Receiving chemotherapy, radiation treatment or immunosuppression drugs.
* Currently enrolled in any other study which may impact on the results of the present study.
* If female: pregnancy, breast-feeding, not currently using and not willing to use an effective form of contraception for 12 months post-surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to healing | 2 weeks, 8 weeks, 12 weeks,16 weeks, 20 weeks, 26 weeks, 39 weeks
  Healing will be assessed both clinically and radiologically (RUST score)

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds General Infirmary, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No